CLINICAL TRIAL: NCT06077318
Title: Comparison of the Sugarbaker and Keyhole Repair for Parastomal Hernia: 10 Years of Experience From a Single Center in China
Brief Title: Comparison of the Sugarbaker and Keyhole Repair for Parastomal Hernia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: Huadong hernia
Record Dates: First submitted 2023-09-19; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia; Keyhole; Sugarbaker; mesh

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Keyhole repair: The keyhole technique involves placing a mesh with a slit in the central hole around the intestinal ring, allowing facilitating the passage of the intestine through the central slit.
  Interventions: Other: Keyhole repair
- Sugarbaker repair: The modified Sugarbaker technique uses a mesh to place a patch on the lateralized intestine, effectively preventing herniation of abdominal contents through the stoma.
  Interventions: Other: Sugarbaker repair

INTERVENTIONS:
Other: Keyhole repair — The keyhole technique involves placing a mesh with a slit in the central hole around the intestinal ring, allowing facilitating the passage of the intestine through the central slit.
  Groups: Keyhole repair
Other: Sugarbaker repair — The modified Sugarbaker technique uses a mesh to place a patch on the lateralized intestine, effectively preventing herniation of abdominal contents through the stoma.
  Groups: Sugarbaker repair

SUMMARY:
Parastomal hernia (PSH) is difficult to manage, with high rates of post-operative recurrence and complication. Keyhole and Sugarbaker are the most commonly used techniques in the surgical repair of the PSH. However, the efficacy and safety of the two surgical methods have not been adequately compared in the East Asian population.

Patients diagnosed with PSH who underwent Sugarbaker or Keyhole repair from August 2012 to August 2022 will be included. Patient demographic data and postoperative outcomes will be retrospectively analyzed. The primary outcome measure is the recurrence rate at one year follow-up time.

DETAILED DESCRIPTION:
Consecutive patients undergoing surgical PSH repair in the Hernia Center of Huadong Hospital Affiliated to Fudan University from August 2012 to August 2022 were included in this study. Huadong Hospital undertakes surgical treatment of complex hernia and abdominal wall diseases in Shanghai, China. The surgical records and clinical data of patients will be retrospectively analyzed. Due to the retrospective design of the study, the patient's informed consent was waived. The study was conducted following the ethical standards set out in the 1964 Declaration of Helsinki and its later amendments.

The patient's surgical strategy was made by the center's experienced colorectal surgeons or specialists in the department of hernia and abdominal wall surgery. In surgical practice, preference is given to the laparoscopic approach, while open surgery is chosen in cases of severe abdominal adhesions. The following three aspects of clinical data were recorded: (1) patients' demographic data, such as age, sex, the primary disease for the stoma, body mass index and comorbidities; (2) Surgical details: repair technique, size of abdominal wall defect, duration of the surgical procedure; (3) Short-term and long-term postoperative outcomes: the primary outcome is the recurrence rate at one year follow-up time, while the secondary outcomes were length and cost of the hospitalization, and rates of the intensive care unit admission, chronic pain, surgical site infection (SSI), re-admission and re-operation rates within 30 days after surgery, major complications after surgery, and surgery-related death.

Only PSH patients who received intraperitoneal onlay Sugarbaker and Keyhole mesh were included. These patients were scheduled for follow-up appointments at the outpatient clinics, specifically at 1 month, 3 months, and 1 year after surgery. If recurrence is suspected by the surgeon after a physical examination, the patient would be requested for an abdominal CT scan. During the CT scan, patients were asked to perform the Valsava maneuver to facilitate the identification of any potential recurrences through imaging. Postoperative major complications were defined as complications requiring hospitalization after surgery to the one-year follow-up time. Patients with follow-up periods of less than one year were excluded from the cohort. Recorded death, recurrence, or loss to follow-up were considered to be the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Only PSH patients who received intraperitoneal onlay Sugarbaker and Keyhole mesh were included.

Exclusion Criteria:

* Patients with less than one year follow-up periods were excluded from the cohort.

Patients received other repair approaches.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with PSH who underwent Sugarbaker or Keyhole repair from August 2012 to August 2022 were included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | one year follow-up time
  recurrence was determined by CT scan

SECONDARY OUTCOMES:
surgical site infection | 30 days after surgery
  wound infection in the surgical site
reoperation and readmission | 30 days after surgery
  rates of the patients suffered from reoperation and readmission
chronic pain | one year follow-up time
  rate of patients suffered from chronic pain in the surgical site
major complication | one year follow-up time
  rate of patients suffered from severe complications (need hospitalization)

REFERENCES:
- [Derived] Shi H, Li S, Lin Y, Yang D, Dong W, Song Z, Song H, Gu Y. Comparison of the 3-D mesh and Sugarbaker repair for parastomal hernia: a single center experience in China. Updates Surg. 2024 Sep;76(5):1991-1996. doi: 10.1007/s13304-024-01946-9. Epub 2024 Jul 21. PMID 39033484